CLINICAL TRIAL: NCT02124993
Title: The Effect of Sleeve Gastrectomy on Food Preference
Acronym: FPQ
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 13029
Record Dates: First submitted 2014-04-22; First posted 2014-04-29 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Severe Obesity
Keywords: Gastrectomy
MeSH Terms: conditions — Obesity, Morbid | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sleeve gastrectomy surgery Participants: Male or female who will undergo a sleeve gastrectomy for obesity by Dr. Drake Bellanger.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Dr. Ballanger's office will administer a FPQ upon approval of an informed consent. Subjects will be asked to complete the questionnaire at a pre-operative visit and six weeks post-operatively.
  Other Names: Food Preference questionnaire (FPQ)

SUMMARY:
This is a questionnaire asking about the sleeve gastrectomy surgery and how has it altered food preferences before and after surgery.

DETAILED DESCRIPTION:
Participants that will undergo the sleeve gastrectomy surgery by Dr. Drake Bellanger's, will be asked to participant in a questionnaire survey. Once given the consent to participate, a food preference questionnaire (FPQ) will be administered at a pre-operative visit and then a six-week follow up visit at Dr. Drake Bellanger's office.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 18 years or over, who will undergo a sleeve gastrectomy for obesity by Dr. Drake Bellanger.

Exclusion Criteria:

* Women who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dr. Drake Bellanger sleeve gastrectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Participants food preferences before sleeve gastrectomy surgery and after surgery. | Change from Baseline in preferences after follow-up six weeks
  A list of food items are on a questionnaire asking food preferences, Breads, Cereals, Grain products, Fruits and Juices, Fats and oils, Milk, etc. which allows the subjects to select their food preferences before and after the surgery.

SECONDARY OUTCOMES:
Participants weight change before sleeve gastrectomy surgery and after surgery focusing on specific macronutrient. | Change from Baseline in weight after follow-up six weeks
  A participant is weighted at baseline visit and follow-up visit 6 weeks after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Greenway, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Dr. Drake Bellanger, Baton Rouge, Louisiana, United States